CLINICAL TRIAL: NCT01207440
Title: A Pivotal Phase 2 Trial of Ponatinib (AP24534) in Patients With Refractory Chronic Myeloid Leukemia and Ph+ Acute Lymphoblastic Leukemia
Brief Title: Ponatinib for Chronic Myeloid Leukemia (CML) Evaluation and Ph+ Acute Lymphoblastic Leukemia (ALL)
Acronym: PACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-10-201; 2010-020414-28 (EudraCT Number)
Record Dates: First submitted 2010-09-20; First posted 2010-09-23 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Chronic Myeloid Leukemia; Ph+ Acute Lymphoblastic Leukemia
Keywords: CML; ALL; PH; ponatinib; Ph+ALL; T315I mutation; Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort A: CP-CML R-I (Experimental): CP-CML participants R-I to dasatinib or nilotinib were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib
- Cohort B: CP-CML with T315I Mutation (Experimental): CP-CML participants who had T315I mutation of breakpoint cluster region-Abelson complex (BCR-ABL) were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib
- Cohort C: Accelerated Phase (AP)-CML R-I (Experimental): AP-CML R-I to dasatinib or nilotinib were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib
- Cohort D: AP-CML with T315I Mutation (Experimental): AP-CML participants who had T315I mutation of BCR-ABL were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib
- Cohort E: Blast Phase (BP)-CML/Ph+ ALL R-I (Experimental): BP-CML or Ph+ ALL R-I to dasatinib or nilotinib or Ph+ ALL R-I to dasatinib or nilotinib were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib
- Cohort F: BP-CML or Ph+ ALL with T315I Mutation (Experimental): BP-CML or Ph+ ALL participants who had T315I mutation of BCR-ABL were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib
- Unassigned to Cohorts A-F (Experimental): Participants who were not assigned to any of the cohorts and have no T315I mutation at study entry and were not R-I to dasatinib or nilotinib, administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib tablets.
  Other Names: AP24534; Iclusig

SUMMARY:
The purpose of this study is to determine the efficacy of ponatinib in patients with chronic myeloid leukemia (CML) in chronic phase (CP), accelerated phase (AP) or blast phase (BP) or with philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia (ALL) who either are resistant or intolerant to either dasatinib or nilotinib, or have the (T)hreonine-315-(I)soleucine (T315I) mutation.

DETAILED DESCRIPTION:
The preliminary analysis of the phase 1 clinical trial revealed evidence of clinical antitumor activity in patients with resistance to approved second-generation tyrosine kinase inhibitors (TKI), dasatinib and nilotinib, including patients with the T315I mutation of the BCR-ABL gene (BCR-ABL). This Phase 1 study, taken together with the strong preclinical data that characterize ponatinib, provides the rationale for moving to a pivotal phase 2 trial of this agent in a population of patients with chronic myeloid leukemia (CML) and Ph+ Acute Lymphoblastic Leukemia (ALL) who are resistant or intolerant to prior TKI therapy and in those patients with the T315I mutation.

PACE is a multi-center, international, phase 2, uncontrolled, open-label trial of oral ponatinib in patients with Philadelphia chromosome-positive (Ph+) disease. The study enrolled 449 patients. Participants assigned to 1 of 6 cohorts in accordance with disease group and received:

* Ponatinib 45 mg

This multi-center trial is conducted worldwide. The overall time to participate in this study is 96 months after last dose of study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have CML in any phase (CP, AP, or BP of any phenotype) or Ph+ ALL
* Previously treated with and developed resistance or intolerance to dasatinib or nilotinib OR developed the T3151 mutation after any tyrosine kinase inhibitor (TKI) therapy
* ≥18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Minimum life expectancy of ≥3 months
* Adequate kidney function
* Adequate liver function
* Normal pancreatic function
* Normal QT Fridericia-corrected interval (QTcF) ≤450 ms for males and ≤470 ms for females
* Negative pregnancy test (if woman of childbearing potential)
* Agree to use effective form of contraception (as applicable)
* Ability to comply with study procedures, in the Investigator's opinion

Exclusion Criteria:

* Received prior TKI treatment within 7 days prior to receiving the first dose of ponatinib, or have not recovered from adverse events (except alopecia) due to agents previously administered.
* Received other therapies as follows:

  1. For CML chronic phase (CP) and accelerated phase (AP) participants, received hydroxyurea or anagrelide within 24 hours prior to receiving the first dose of ponatinib; interferon, cytarabine, or immunotherapy within 14 days prior to first dose of ponatinib; or any other cytotoxic chemotherapy, radiotherapy, or investigational therapy within 28 days prior to receiving the first dose of ponatinib.
  2. For CML blast phase (BP) participants, received chemotherapy within 14 days prior to the first dose of ponatinib.
  3. For Ph+ ALL participants, received corticosteroids within 24 hours before the first dose of ponatinib; or vincristine within 7 days prior to the first dose of ponatinib; or received other chemotherapy within 14 days prior to the first dose of ponatinib.
* Underwent stem cell transplant <60 days prior to receiving first dose of ponatinib
* Evidence of on-going graft versus-host disease (GVHD), or GVHD requiring immunosuppressive therapy
* Taking medications that are known to be associated with Torsades de Pointes
* Require concurrent treatment with immunosuppressive agents (other than corticosteroids prescribed for a short course of therapy)
* Previously treated with ponatinib
* CML CP participants are excluded if they are in Complete cytogenetic response (CCyR)
* Participants with CML AP, CML BP, or Ph+ ALL are excluded if they are in Major Hematologic Response (MaHR).
* Have active Central Nervous System (CNS) disease
* Have significant or active cardiovascular disease
* Have a significant bleeding disorder unrelated to CML or Ph+ALL
* Have a history of pancreatitis or alcohol abuse
* Have uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL)
* Have malabsorption syndrome or other gastrointestinal illness that could affect absorption of ponatinib
* Diagnosed with another primary malignancy in the past 3 years
* Pregnant or lactating
* Underwent major surgery within 14 days prior to first dose of ponatinib
* Have ongoing or active infection
* Suffer from any other condition or illness that would compromise safety or interfere with evaluation of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (42):
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
- Belgium (2):
  - UCL Bruxelles, Brussels
  - UZ Leuven, Leuven
- France (9):
  - Institut Bergonie, Bordeaux
  - Hopital Andre Mignot, Le Chesnay
  - Hopital Claude Huriez CHRU, Lille
  - Chu Brabois, Nancy
  - Hopital Archet, Nice
  - Hopital St. Louis, Paris
  - Hopital Edouard Herriot, Pierre-Bénite
  - Entre Hospitalier Universitaire, Poitiers
  - Hopital de Purpan, Toulouse
- Germany (5):
  - Charite - Universitatsmedizin Berlin,, Berlin
  - Klinikum der Goethe Universitat,, Frankfurt
  - Universitatsklinikum Jena, Jena
  - University of Heidelberg, Mannheim
  - III. Med. Klinik und Poliklinik, München
- Italy (5):
  - Universita di Bologna, Bologna
  - University of Modena, Modena
  - University of Milano Bicocca, Monza
  - University of Turin, Orbassano (TO)
  - University Tor Vergata, Roma
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groeningen, Groningen
- Singapore General Hospital, Singapore, Singapore
- The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, South Korea
- Spain (4):
  - Hospital Clinic, Barcelona
  - La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clinico of Valencia, Valencia
- Sweden (3):
  - Lund University, Lund
  - Karolinska Hospital, Stockholm
  - University Hospital Uppsala, Uppsala
- United Kingdom (5):
  - Gartnavel General Hospital, Glasgow
  - Royal Liverpool University Hospital, Liverpool
  - Hammersmith Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Cortes JE, Kim DW, Pinilla-Ibarz J, le Coutre PD, Paquette R, Chuah C, Nicolini FE, Apperley JF, Khoury HJ, Talpaz M, DeAngelo DJ, Abruzzese E, Rea D, Baccarani M, Muller MC, Gambacorti-Passerini C, Lustgarten S, Rivera VM, Haluska FG, Guilhot F, Deininger MW, Hochhaus A, Hughes TP, Shah NP, Kantarjian HM. Ponatinib efficacy and safety in Philadelphia chromosome-positive leukemia: final 5-year results of the phase 2 PACE trial. Blood. 2018 Jul 26;132(4):393-404. doi: 10.1182/blood-2016-09-739086. Epub 2018 Mar 22. PMID 29567798
- [Derived] Kantarjian HM, Jabbour E, Deininger M, Abruzzese E, Apperley J, Cortes J, Chuah C, DeAngelo DJ, DiPersio J, Hochhaus A, Lipton J, Nicolini FE, Pinilla-Ibarz J, Rea D, Rosti G, Rousselot P, Shah NP, Talpaz M, Srivastava S, Ren X, Mauro M. Ponatinib after failure of second-generation tyrosine kinase inhibitor in resistant chronic-phase chronic myeloid leukemia. Am J Hematol. 2022 Nov;97(11):1419-1426. doi: 10.1002/ajh.26686. Epub 2022 Aug 30. PMID 36054756
- [Derived] Januzzi JL, Garasic JM, Kasner SE, McDonald V, Petrie MC, Seltzer J, Mauro M, Croce K, Berman E, Deininger M, Hochhaus A, Pinilla-Ibarz J, Nicolini F, Kim DW, DeAngelo DJ, Kantarjian H, Xu J, Hall T, Srivastava S, Naranjo D, Cortes J. Retrospective analysis of arterial occlusive events in the PACE trial by an independent adjudication committee. J Hematol Oncol. 2022 Jan 6;15(1):1. doi: 10.1186/s13045-021-01221-z. PMID 34991679
- [Derived] Cortes JE, Kim DW, Pinilla-Ibarz J, le Coutre P, Paquette R, Chuah C, Nicolini FE, Apperley JF, Khoury HJ, Talpaz M, DiPersio J, DeAngelo DJ, Abruzzese E, Rea D, Baccarani M, Muller MC, Gambacorti-Passerini C, Wong S, Lustgarten S, Rivera VM, Clackson T, Turner CD, Haluska FG, Guilhot F, Deininger MW, Hochhaus A, Hughes T, Goldman JM, Shah NP, Kantarjian H; PACE Investigators. A phase 2 trial of ponatinib in Philadelphia chromosome-positive leukemias. N Engl J Med. 2013 Nov 7;369(19):1783-96. doi: 10.1056/NEJMoa1306494. Epub 2013 Nov 1. PMID 24180494
- [Derived] O'Hare T, Zabriskie MS, Eiring AM, Deininger MW. Pushing the limits of targeted therapy in chronic myeloid leukaemia. Nat Rev Cancer. 2012 Jul 24;12(8):513-26. doi: 10.1038/nrc3317. PMID 22825216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 66 investigative sites in the Australia, Belgium, Canada, France, Germany, Italy, the Netherlands, Republic of Korea, Singapore, Spain, Sweden, the United Kingdom and the United States from 30 September 2010 to 17 January 2019.
Pre-assignment Details: Participants were assigned to 1 of 6 cohorts: chronic myeloid leukemia (CML) in chronic (CP), accelerated (AP), or blast phase (BP), or with Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ALL) who were resistant or intolerant (R-I) to either dasatinib or nilotinib or had (T)hreonine-315-(I)soleucine (T315I) mutation.
Groups:
- Cohort C: AP-CML R-I: AP-CML R-I to dasatinib or nilotinib were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
- Cohort E: BP-CML/Ph+ ALL R-I: BP-CML or Ph+ ALL R-I to dasatinib or nilotinib or Ph+ ALL R-I to dasatinib or nilotinib were administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
- Unassigned to Cohorts A-F: Participants who were not assigned to any of the cohorts and have no T315I mutation at study entry and were not resistant or intolerant to dasatinib or nilotinib, administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
Period: Overall Study
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation | Unassigned to Cohorts A-F
Started | 203 | 64 | 65 | 18 | 48 | 46 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 203 | 64 | 65 | 18 | 48 | 46 | 5
Not completed — Adverse Event | 46 | 11 | 7 | 2 | 6 | 6 | 2
Not completed — Death | 6 | 3 | 2 | 2 | 7 | 5 | 1
Not completed — Lack of Efficacy | 13 | 2 | 5 | 1 | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 5 | 5 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 19 | 10 | 19 | 7 | 23 | 27 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 69 | 19 | 12 | 2 | 3 | 0 | 2
Not completed — Withdrawal by Subject | 29 | 4 | 5 | 3 | 2 | 2 | 0
Not completed — Reason Not Specified | 10 | 10 | 7 | 0 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of ponatinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation | Unassigned to Cohorts A-F | Total
Number analyzed (Participants) | 203 | 64 | 65 | 18 | 48 | 46 | 5 | 449
Age, Continuous [Median (Full Range); unit: years] | 61.0 [22 to 94] | 52.0 [18 to 87] | 60.0 [23 to 82] | 54.0 [24 to 78] | 54.0 [18 to 74] | 56.0 [18 to 80] | 63.0 [51 to 71] | 59.0 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 16 | 40 | 7 | 17 | 20 | 3 | 211
  Male | 95 | 48 | 25 | 11 | 31 | 26 | 2 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 6 | 1 | 2 | 12 | 0 | 42
  Not Hispanic or Latino | 190 | 56 | 59 | 17 | 46 | 34 | 5 | 407
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska native | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 17 | 14 | 8 | 3 | 8 | 7 | 2 | 59
  Black/African American | 7 | 4 | 7 | 5 | 1 | 1 | 0 | 25
  White | 174 | 42 | 47 | 9 | 39 | 38 | 3 | 352
  Unknown | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 8
  Other | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG-PS measured on-therapy assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hrs), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Population: 1 participant from the cohort F had missing ECOG data.
  Participants
    number analyzed (Participants) | 203 | 64 | 65 | 18 | 47 | 46 | 5 | 448
    ECOG=0 | 139 | 47 | 33 | 12 | 15 | 16 | 5 | 267
    ECOG=1 | 60 | 17 | 25 | 6 | 20 | 19 | 0 | 147
    ECOG=2 | 4 | 0 | 7 | 0 | 12 | 11 | 0 | 34
Time From Diagnosis to First Dose [Median (Full Range); unit: years] | 7.85 [0.45 to 27.43] | 4.78 [1.16 to 19.49] | 7.13 [0.33 to 28.47] | 6.61 [1.17 to 15.90] | 3.96 [0.62 to 27.21] | 1.63 [0.46 to 14.14] | 4.80 [1.74 to 18.60] | 6.09 [0.33 to 28.47]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of CP-CML Participants With Major Cytogenetic Response (MCyR)
Description: MCyR is defined as percentage of participants with complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). Cytogenetic response is the percentage of Philadelphia chromosome positive (Ph+) metaphases in bone marrow (BM). Response is further defined as MCyR: CCyR or PCyR, where CCyR: no Ph+ cells; PCyR: 1 to 35% Ph+ cells.
Time Frame: Up to 12 months after initiation of study treatment
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib. The data for this outcome measure is applicable for Cohorts A and B only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation
Number analyzed (Participants) | 203 | 64
percentage of participants | 50.7 [43.6 to 57.8] | 70.3 [57.6 to 81.1]

2. Primary Outcome: Percentage of AP-CML Participants With Major Hematologic Response (MaHR)
Description: MaHR is defined as percentage of participants with complete hematologic response (CHR) or no evidence of leukemia (NEL). Response criteria for CHR is reported as white blood cells (WBC)≤institutional upper limit of normal, absolute neutrophil count (ANC)≥1000/mm^3, platelets≥100,000/mm^3, no blasts or promyelocytes in peripheral blood, BM blasts ≤5%, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement; Response criteria for NEL is reported as WBC≤institutional upper limit of normal, no blasts or promyelocytes in peripheral blood, BM blasts ≤5%, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement, at least 1 of the following: (i) 20,000/mm^3≤platelets<100,000/mm^3; (ii) 500/mm^3≤ANC<1000/mm^3.
Time Frame: Up to 6 months after initiation of study treatment
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib. The data for this outcome measure is applicable for Cohorts C and D only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation
Number analyzed (Participants) | 65 | 18
percentage of participants | 56.9 [44.0 to 69.2] | 55.6 [30.8 to 78.5]

3. Primary Outcome: Percentage of BP-CML/Ph+ ALL Participants With MaHR
Description: MaHR is defined as percentage of participants with CHR or NEL. Response criteria for CHR is reported as WBC≤institutional upper limit of normal, ANC≥1000/mm^3, platelets ≥100,000/mm^3, no blasts or promyelocytes in peripheral blood, BM blasts ≤5%, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement; Response criteria for NEL is reported as WBC≤ institutional upper limit of normal, no blasts or promyelocytes in peripheral blood, BM blasts ≤5%, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement, at least 1 of the following: (i) 20,000/mm^3 ≤platelets<100,000/mm^3; (ii) 500/mm^3≤ANC<1000/mm^3.
Time Frame: Up to 6 months after initiation of study treatment
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib. The data for this outcome measure is applicable for Cohorts E and F only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 48 | 46
percentage of participants | 35.4 [22.2 to 50.5] | 32.6 [19.5 to 48.0]

4. Secondary Outcome: Percentage of CP-CML Participants With CHR
Description: Response criteria for CHR is reported as WBC≤institutional upper limit of normal, platelets<450,000/mm^3, no blasts or promyelocytes in peripheral blood, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, no extramedullary involvement (including no hepatomegaly or splenomegaly).
Time Frame: Every 3 cycles up to 39 cycles, followed by every subsequent sixth cycle (Up to approximately 48 months after first dose)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation
Number analyzed (Participants) | 203 | 64
percentage of participants | 94.6 [90.5 to 97.3] | 92.2 [82.7 to 97.4]

5. Secondary Outcome: Percentage of CP-CML Participants With Confirmed MCyR
Description: Confirmed MCyR is defined as 2 assessments of CCyR or PCyR at least 28 days apart. For CP participants entering the trial in PCyR, confirmed MCyR is defined as 2 assessments of CCyR at least 28 days apart.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation
Number analyzed (Participants) | 203 | 64
percentage of participants | 40.9 [34.1 to 48.0] | 62.5 [49.5 to 74.3]

6. Secondary Outcome: Percentage of CP-CML Participants With Major Molecular Response (MMR)
Description: MMR is defined as a ratio of reverse transcribed transcript of BCR-ABL to ABL ≤0.1% on the international scale (equivalent to a 3-log reduction in transcript).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation
Number analyzed (Participants) | 203 | 64
percentage of participants | 35.0 [28.4 to 42.0] | 57.8 [44.8 to 70.1]

7. Secondary Outcome: Percentage of AP-CML or BP-CML/Ph+ ALL Participants With MCyR
Description: MCyR is defined as percentage of participants with CCyR or PCyR. Cytogenetic response is the percentage of Ph+ metaphases in BM. Response is further defined as MCyR: CCyR or PCyR, where CCyR: no Ph+ cells; PCyR: 1 to 35% Ph+ cells.
Time Frame: Every 2 cycles up to 26 cycles, followed by every 3 cycles from cycles 27 through 39, and then every subsequent sixth cycle (Up to approximately 48 months after first dose)
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib. The data for this outcome measure is applicable for Cohorts C to F only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 65 | 18 | 48 | 46
percentage of participants | 33.8 [22.6 to 46.6] | 55.6 [30.8 to 78.5] | 27.1 [15.3 to 41.8] | 34.8 [21.4 to 50.2]

8. Secondary Outcome: Percentage of AP-CML or BP-CML/Ph+ ALL Participants With Confirmed MCyR
Description: Confirmed MCyR is defined as 2 assessments of CCyR or PCyR at least 28 days apart.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 65 | 18 | 48 | 46
percentage of participants | 24.6 [14.8 to 36.9] | 38.9 [17.3 to 64.3] | 20.8 [10.5 to 35.0] | 15.2 [6.3 to 28.9]

9. Secondary Outcome: Percentage of AP-CML or BP-CML/Ph+ ALL Participants With MMR
Description: as for outcome 6
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 65 | 18 | 48 | 46
percentage of participants | 18.5 [9.9 to 30.0] | 33.3 [13.3 to 59.0] | 18.8 [8.9 to 32.6] | 4.3 [0.5 to 14.8]

10. Secondary Outcome: Time to Response
Description: Time to response is defined as the interval from the first dose of study treatment until the criteria for response are first met, censored at the last assessment of response. Median time to response was estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 48 months after first dose
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib. Median time to response was reported for responders only. Participants who did not achieve the specified response were censored at the last response assessment. Number analyzed: participants with data available at given time-point.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 203 | 64 | 65 | 18 | 48 | 46
days
  Hematologic Response: number analyzed (Participants) | 192 | 59 | 37 | 10 | 17 | 15
  Hematologic Response | 13.0 [1 to 417] | 10.0 [4 to 1008] | 21.0 [12 to 112] | 20.5 [14 to 176] | 28.0 [14 to 168] | 24.0 [11 to 57]
  Cytogenetic Response: number analyzed (Participants) | 103 | 45 | 22 | 10 | 13 | 16
  Cytogenetic Response | 85.0 [56 to 343] | 84.0 [49 to 333] | 113.5 [26 to 280] | 83.0 [25 to 295] | 28.0 [28 to 168] | 56.0 [27 to 112]
  Molecular Response: number analyzed (Participants) | 71 | 37 | 12 | 6 | 9 | 2
  Molecular Response | 173.0 [55 to 1686] | 167.0 [81 to 756] | 340.5 [55 to 1364] | 335.5 [107 to 925] | 56.0 [54 to 113] | 63.0 [59 to 67]

11. Secondary Outcome: Duration of Response
Description: Duration of Response is defined as the interval between the first assessment at which the criteria for response are met until the criteria for progression are met, censored at the last date at which the criteria for response are met. Duration of response was estimated by the Kaplan-Meier method as the probability of remaining in response.
Time Frame: Up to approximately 48 months after first dose
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib. Number analyzed is number of participants with data available for analysis at given time-point
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 203 | 64 | 65 | 18 | 48 | 46
days
  Hematologic Response: number analyzed (Participants) | 192 | 59 | 37 | 10 | 17 | 15
  Hematologic Response | NA [36 to 2172] — Duration of response was not reached for Cohorts A and B due to fewer number of participants with events. | NA [33 to 2171] — Duration of response was not reached for Cohorts A and B due to fewer number of participants with events. | 360.0 [35 to 2079] | 732.0 [42 to 1334] | 196.0 [54 to 1811] | 108.0 [54 to 1038]
  Cytogenetic Response: number analyzed (Participants) | 103 | 45 | 22 | 10 | 13 | 16
  Cytogenetic Response | NA [1 to 1963] — Duration of response was not reached for Cohorts A and B due to fewer number of participants with events. | NA [1 to 1903] — Duration of response was not reached for Cohorts A and B due to fewer number of participants with events. | NA [1 to 1779] — Duration of response was not reached due to fewer number of participants with events. | 728.0 [28 to 1569] | NA [1 to 1770] — Duration of response was not reached due to fewer number of participants with events. | 63.0 [1 to 673]
  Molecular Response: number analyzed (Participants) | 71 | 37 | 12 | 6 | 9 | 2
  Molecular Response | NA [78 to 1891] — Duration of response was not reached for Cohorts A and B due to fewer number of participants with events. | NA [1 to 1899] — Duration of response was not reached for Cohorts A and B due to fewer number of participants with events. | 560.0 [1 to 1666] | 222.0 [1 to 783] | NA [1 to 1742] — Duration of response was not reached due to fewer number of participants with events. | 98.0 [1 to 98]

12. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval from the first dose of study treatment until the criteria for progression or death are met, censored at the last response assessment. Progression from CP is reported as death, development of AP or BP, loss of CHR (in the absence of cytogenetic response), confirmed by development in complete blood counts (CBCs) at least 4 weeks apart, loss of MCyR, increasing WBC in participant without CHR defined by doubling of WBC to >20K on 2 occasions at least 4 weeks apart; Progression from AP is reported as death, development of confirmed BP, loss of previous major or minor hematologic response over a 2-week period, no decrease from baseline levels in percentage blasts in peripheral blood or BM on all assessments over a 4-week period; Progression from BP or Ph+ ALL is reported as death, increasing blasts in peripheral blood or BM over a 4 week period.
Time Frame: Every 12 weeks ± 2 weeks from last dose of study drug or the investigator/participant decision to discontinue treatment, whichever occurred later (Up to approximately 96 months after last dose)
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 203 | 64 | 65 | 18 | 48 | 46
days | NA [1285.0 to NA] — PFS was not reached for Cohorts A and B due to fewer number of participants with events. | 1809.0 [1028.0 to NA] — PFS was not reached for Cohorts A and B due to fewer number of participants with events. | 432.0 [335.0 to 714.0] | 959.0 [186.0 to 1847.0] | 111.0 [55.0 to 169.0] | 83.0 [55.0 to 150.0]

13. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval from the first dose of study treatment until death, censored at the last date at which participant was known to be alive.
Time Frame: From the first dose of study treatment until death (Up to 96 months post last dose)
Population: Treated population included all participants assigned to Cohorts A to F who received at least 1 dose of ponatinib.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation
Number analyzed (Participants) | 203 | 64 | 65 | 18 | 48 | 46
days | NA [NA to NA] — Median OS has not been reached for Cohort A and B due to fewer number of participants with events. | NA [NA to NA] — Median OS has not been reached for Cohort A and B due to fewer number of participants with events. | 1689.0 [969.0 to NA] — Upper limit of 95% confidence interval was not estimable due to fewer number of participants with events. | 1847.0 [281.0 to 2143.0] | 209.0 [119.0 to 379.0] | 200.0 [150.0 to 279.0]

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Event (TEAE) and Serious AE (SAE)
Description: An AE is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent. A TEAE is defined as an AE that occurs after administration of first dose of study drug and through 30 days after last dose of study drug or until start of subsequent antineoplastic therapy.
Time Frame: From first dose up to 30 days after last dose of the study drug (Up to approximately 49 months)
Population: The safety population included all participants who received at least 1 dose of ponatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation | Unassigned to Cohorts A-F
Number analyzed (Participants) | 203 | 64 | 65 | 18 | 48 | 46 | 5
Participants
  TEAE | 203 | 64 | 65 | 18 | 48 | 46 | 5
  SAE | 132 | 39 | 44 | 13 | 41 | 37 | 3

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs: From first dose up to 30 days after last dose of the study drug (Up to approximately 49 months); All-Cause Mortality: Up to approximately 8 years
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Unassigned AP/CP-CML: Participants who were not assigned to any of the cohorts and have no T315I mutation at study entry and were not R-I to dasatinib or nilotinib, administered ponatinib 45 mg, tablet, orally, once daily until disease progression or development of intolerance or if they met one or more of the protocol defined criteria for discontinuation (Up to approximately 48 months).
Arm/Group | Cohort A: CP-CML R-I | Cohort B: CP-CML With T315I Mutation | Cohort C: AP-CML R-I | Cohort D: AP-CML With T315I Mutation | Cohort E: BP-CML/Ph+ ALL R-I | Cohort F: BP-CML or Ph+ ALL With T315I Mutation | Unassigned AP/CP-CML
All-Cause Mortality (participants affected / at risk) | 41/203 | 18/64 | 30/65 | 9/18 | 40/48 | 39/46 | 2/5
Serious Adverse Events (participants affected / at risk) | 132/203 | 39/64 | 44/65 | 13/18 | 41/48 | 37/46 | 3/5
Other Adverse Events (participants affected / at risk) | 203/203 | 64/64 | 65/65 | 18/18 | 48/48 | 46/46 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: CP-CML R-I (N=203) | Cohort B: CP-CML With T315I Mutation (N=64) | Cohort C: AP-CML R-I (N=65) | Cohort D: AP-CML With T315I Mutation (N=18) | Cohort E: BP-CML/Ph+ ALL R-I (N=48) | Cohort F: BP-CML or Ph+ ALL With T315I Mutation (N=46) | Unassigned AP/CP-CML (N=5)
Pancreatitis (Gastrointestinal disorders) | 10 | 4 | 3 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 4 | 1 | 4 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 11 | 4 | 0 | 0 | 3 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 3 | 1 | 0 | 1 | 1 | 0 — Two treatment-emergent deaths (1-Cohort B, 1-Cohort E) occurred during treatment with ponatinib and are not related.
Coronary artery disease (Cardiac disorders) | 4 | 6 | 1 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 1 | 2 | 2 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort A and is related.
Angina pectoris (Cardiac disorders) | 10 | 4 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 — Four treatment-emergent deaths (2-Cohort A, 1-Cohort B, 1-Cohort F) occurred during treatment with ponatinib and one in Cohort F is related.
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 1 | 1 | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 5 | 8 | 1 | 4 | 5 | 0 — Two treatment-emergent deaths occurred during treatment with ponatinib in Cohort A and one is related.
Cellulitis (Infections and infestations) | 4 | 1 | 2 | 1 | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 2 | 1 | 2 | 2 | 1 — Three treatment-emergent deaths (1-Cohort D, 1-Cohort E, 1-Cohort F) occurred during treatment with ponatinib and are not related.
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 2 | 0 | 1 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 4 | 3 | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 0 | 2 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 3 | 5 | 2 | 2 | 2 | 1
Non-cardiac chest pain (General disorders) | 4 | 1 | 2 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 7 | 4 | 14 | 8 | 0 — Twenty-four treatment-emergent deaths (4-Cohort A, 1-Cohort B, 2-Cohort C, 2-Cohort D, 10-Cohort E, 5 Cohort F) occurred during treatment with ponatinib and are not related.
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 11 | 0 | 2 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort C and is not related.
Deep vein thrombosis (Vascular disorders) | 4 | 1 | 0 | 0 | 1 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort F and is not related.
Cerebrovascular accident (Nervous system disorders) | 5 | 4 | 1 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort B and is not related.
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral artery stenosis (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 5 | 3 | 0 | 0 | 0 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort B and is not related.
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
IVth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 0 | 4 | 0 | 2 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 5 | 5 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 1 | 0 | 2 | 1 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort E and is not related.
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 0 | 2 | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort D and is related.
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 — Three treatment-emergent deaths (1-Cohort C, 2-Cohort F) occurred during treatment with ponatinib and are not related.
Splenic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 1 | 0 — Three treatment-emergent deaths (1-Cohort C, 1-Cohort E, 1-Cohort F) occurred during treatment with ponatinib and are not related.
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 2 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort F and is not related.
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort F and is not related.
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort F and is not related.
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort E and is not related.
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 — One treatment-emergent death occurred during treatment with ponatinib in Unassigned AP/CP-CML and is related.
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort E and is related.
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Implant site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort E and is not related.
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cardiac Discomfort (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dressler's syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis Noninfective (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort E and is related.
Impaired healing (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular stent occlusion (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 — Two treatment-emergent deaths (1-Cohort E, 1-Cohort F) occurred during treatment with ponatinib and are not related.
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Genital infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Iiird nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort E and is not related.
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 2 | 0 | 3 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort A and is not related.
Large cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort D and is not related.
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucocutaneous haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 10 | 4 | 1 | 1 | 1 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 4 | 3 | 0 | 0 | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 4 | 1 | 0 | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Dry gangrene (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Coeliac artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immobile (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 0 | 2 | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 4 | 2 | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 5 | 1 | 2 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
JC polyomavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with ponatinib in Cohort A and is not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: CP-CML R-I (N=203) | Cohort B: CP-CML With T315I Mutation (N=64) | Cohort C: AP-CML R-I (N=65) | Cohort D: AP-CML With T315I Mutation (N=18) | Cohort E: BP-CML/Ph+ ALL R-I (N=48) | Cohort F: BP-CML or Ph+ ALL With T315I Mutation (N=46) | Unassigned AP/CP-CML (N=5)
Anaemia (Blood and lymphatic system disorders) | 39 | 7 | 20 | 7 | 14 | 11 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0 | 3 | 3 | 0
Hypochromasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 0 | 5 | 2 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 6 | 0 | 2 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 42 | 6 | 24 | 4 | 13 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 90 | 18 | 32 | 4 | 16 | 7 | 1
Angina pectoris (Cardiac disorders) | 9 | 4 | 3 | 0 | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 3 | 1 | 0 | 2 | 4 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Palpitations (Cardiac disorders) | 6 | 1 | 2 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 5 | 1 | 2 | 0 | 3 | 2 | 0
Tachycardia (Cardiac disorders) | 3 | 1 | 1 | 0 | 2 | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 8 | 1 | 1 | 1 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 8 | 1 | 3 | 1 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 7 | 2 | 4 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 7 | 1 | 1 | 1 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 16 | 5 | 4 | 2 | 4 | 3 | 1
Eye pain (Eye disorders) | 8 | 4 | 2 | 0 | 3 | 0 | 0
Eyelid disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 13 | 6 | 3 | 1 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 8 | 3 | 3 | 0 | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 12 | 7 | 4 | 1 | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 75 | 21 | 20 | 7 | 7 | 10 | 2
Abdominal pain upper (Gastrointestinal disorders) | 40 | 10 | 11 | 2 | 6 | 8 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 89 | 21 | 16 | 7 | 21 | 13 | 3
Dental necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 43 | 10 | 17 | 7 | 15 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 20 | 6 | 4 | 0 | 4 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 12 | 6 | 4 | 0 | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 8 | 2 | 0 | 2 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 2 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 1 | 1 | 1 | 2 | 2 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 53 | 24 | 22 | 5 | 16 | 12 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 11 | 2 | 4 | 1 | 2 | 3 | 0
Toothache (Gastrointestinal disorders) | 13 | 0 | 3 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 38 | 12 | 17 | 6 | 14 | 11 | 0
Asthenia (General disorders) | 40 | 8 | 5 | 4 | 3 | 8 | 0
Chest pain (General disorders) | 13 | 4 | 1 | 1 | 1 | 0 | 1
Chills (General disorders) | 16 | 4 | 6 | 4 | 7 | 2 | 1
Fatigue (General disorders) | 60 | 21 | 22 | 8 | 16 | 9 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 10 | 3 | 4 | 0 | 1 | 1 | 0
Localised oedema (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 13 | 6 | 3 | 0 | 2 | 2 | 0
Oedema peripheral (General disorders) | 36 | 8 | 9 | 5 | 12 | 5 | 1
Pain (General disorders) | 19 | 7 | 8 | 3 | 8 | 3 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 5 | 4 | 5 | 2 | 0 | 1 | 0
Pyrexia (General disorders) | 52 | 13 | 20 | 11 | 16 | 12 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 1 | 2 | 1 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 2 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 19 | 5 | 3 | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 6 | 1 | 4 | 1 | 4 | 2 | 0
Conjunctivitis (Infections and infestations) | 9 | 2 | 2 | 2 | 0 | 0 | 1
Cystitis (Infections and infestations) | 5 | 0 | 1 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 8 | 6 | 3 | 1 | 1 | 2 | 1
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 1 | 2 | 1 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 11 | 1 | 2 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 4 | 1 | 0 | 1 | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 26 | 7 | 9 | 5 | 1 | 2 | 1
Oral candidiasis (Infections and infestations) | 4 | 1 | 1 | 1 | 3 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 1 | 2 | 1 | 4 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 17 | 7 | 3 | 0 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 4 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 2 | 1 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 6 | 0 | 4 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 16 | 18 | 9 | 2 | 6 | 2 | 1
Urinary tract infection (Infections and infestations) | 18 | 5 | 9 | 3 | 2 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 1 | 1 | 0 | 3 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 1 | 1 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 2 | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 2 | 1 | 0
Transfusion related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 39 | 12 | 15 | 4 | 7 | 5 | 0
Amylase increased (Investigations) | 19 | 2 | 6 | 1 | 4 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 31 | 11 | 11 | 5 | 7 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 20 | 5 | 9 | 0 | 3 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 4 | 1 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 9 | 3 | 1 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 8 | 4 | 5 | 0 | 5 | 1 | 0
Blood glucose increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 6 | 2 | 1 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 16 | 5 | 5 | 3 | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 56 | 15 | 10 | 2 | 8 | 3 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 8 | 2 | 0 | 3 | 5 | 2 | 0
Platelet count decreased (Investigations) | 15 | 3 | 6 | 1 | 2 | 3 | 0
Platelet count increased (Investigations) | 3 | 1 | 1 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 23 | 5 | 7 | 0 | 5 | 2 | 1
White blood cell count decreased (Investigations) | 4 | 1 | 2 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 28 | 7 | 10 | 2 | 7 | 8 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 4 | 1 | 1 | 3 | 0 | 0
Gout (Metabolism and nutrition disorders) | 3 | 5 | 1 | 1 | 3 | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 4 | 2 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 7 | 9 | 0 | 3 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3 | 1 | 2 | 5 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 16 | 3 | 3 | 2 | 5 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 1 | 8 | 1 | 5 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 4 | 3 | 2 | 11 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 0 | 3 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 2 | 3 | 2 | 2 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 10 | 3 | 3 | 1 | 5 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 72 | 18 | 22 | 6 | 10 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 8 | 10 | 3 | 8 | 7 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 32 | 6 | 8 | 3 | 8 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 32 | 6 | 4 | 1 | 3 | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 0 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 | 5 | 4 | 2 | 3 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 18 | 14 | 4 | 10 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 13 | 1 | 3 | 0 | 2 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 56 | 9 | 11 | 5 | 6 | 6 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 34 | 12 | 7 | 2 | 4 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 6 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 87 | 27 | 18 | 7 | 15 | 12 | 1
Hypoaesthesia (Nervous system disorders) | 11 | 2 | 1 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 6 | 0 | 1 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 15 | 1 | 2 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 15 | 5 | 1 | 1 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 11 | 0 | 4 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Vith nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 10 | 3 | 11 | 4 | 4 | 3 | 0
Confusional state (Psychiatric disorders) | 4 | 1 | 1 | 2 | 2 | 3 | 0
Depression (Psychiatric disorders) | 13 | 2 | 5 | 0 | 3 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 25 | 5 | 10 | 1 | 10 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 1 | 0 | 3 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 6 | 2 | 3 | 2 | 3 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 7 | 0 | 1 | 0 | 3 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 4 | 1 | 2 | 1 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 4 | 1 | 3 | 1 | 0 | 2 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 9 | 6 | 4 | 4 | 1 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 11 | 15 | 3 | 8 | 6 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 14 | 12 | 4 | 11 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 3 | 6 | 1 | 5 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 4 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 4 | 3 | 8 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 7 | 2 | 8 | 4 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2 | 1 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 4 | 5 | 4 | 4 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 84 | 28 | 21 | 4 | 15 | 9 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 0 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 22 | 6 | 6 | 1 | 3 | 4 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 4 | 0 | 0 | 1 | 2
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 17 | 7 | 4 | 1 | 1 | 3 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 15 | 10 | 4 | 1 | 2 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 6 | 6 | 1 | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 28 | 3 | 10 | 3 | 2 | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 39 | 21 | 9 | 2 | 11 | 8 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 9 | 4 | 0 | 1 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 11 | 4 | 1 | 3 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 14 | 4 | 5 | 1 | 3 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 21 | 6 | 5 | 3 | 2 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 12 | 6 | 2 | 1 | 0 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 1 | 3 | 1 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 0
Activities of daily living impaired (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 8 | 2 | 4 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 12 | 1 | 4 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 68 | 21 | 13 | 8 | 13 | 8 | 2
Hypotension (Vascular disorders) | 6 | 0 | 1 | 0 | 3 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2010-12-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT01207440/SAP_000.pdf
  • Study Protocol (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT01207440/Prot_001.pdf